CLINICAL TRIAL: NCT02779114
Title: A Phase 3, Multicenter, Randomized, Open, Prospective, Controlled, Parallel Group Study of Reduction of Therapy in Patients With Rheumatoid Arthritis in Ongoing Remission.
Brief Title: RETRO (REduction of Therapy in RA Patients in Ongoing Remission)
Acronym: RETRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKER00109STUM3
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Remission; Dose reduction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Other): After 1:1:1 randomization patients in the control group receive their previous disease modifying therapy of conventional DMARD, biologicals and glucocorticoids during 12 months of the study.
  Interventions: Drug: Control group; Other: Reduction group 1; Other: Reduction group 2
- Reduction group 1 (Other): Patients in reduction group 1 receive exactly 50% of their previous disease modifying therapy of conventional DMARD, biologicals and glucocorticoids during the first six months of the study.
  Interventions: Drug: Control group; Other: Reduction group 1; Other: Reduction group 2
- Reduction group 2 (Other): Patients in reduction group 2 receive exactly 50% of their previous disease modifying therapy of conventional DMARD, biologicals and glucocorticoids during the first six months of the study. If they are still in remission they will discontinue their previous disease modifying therapy of conventional DMARD, biologicals and glucocorticoids during the first six months of the study.
  Interventions: Drug: Control group; Other: Reduction group 1; Other: Reduction group 2

INTERVENTIONS:
Drug: Control group — Stable dosage of previous treatment with Decortin H®, Leflunomid (e.g. Arava®), Ciclosporin (e.g. Immunosporin®), Sulfasalazin (e.g. Azulfidine RA®, Pleon RA®), Hydroxychloroquine (e.g. Quensyl®); Azathioprin, Methotrexate (e.g. Lantarel®, Metex®), Etanercept (Enbrel®), Adalimumab (Humira®), Infliximab (Remicade®), Tocilizumab (RoActemra®), Golimumab (Simponi®), Certolizumab (Cimzia®), Abatacept (Orencia®)
Other: Reduction group 1 — Dose reduction of 50% for 12 months of previous treatment with Decortin H®, Leflunomid (e.g. Arava®), Ciclosporin (e.g. Immunosporin®), Sulfasalazin (e.g. Azulfidine RA®, Pleon RA®), Hydroxychloroquine (e.g. Quensyl®); Azathioprin, Methotrexate (e.g. Lantarel®, Metex®), Etanercept (Enbrel®), Adalimumab (Humira®), Infliximab (Remicade®), Tocilizumab (RoActemra®), Golimumab (Simponi®), Certolizumab (Cimzia®), Abatacept (Orencia®)
Other: Reduction group 2 — Dose reduction of 50% of previous treatment with Decortin H®, Leflunomid (e.g. Arava®), Ciclosporin (e.g. Immunosporin®), Sulfasalazin (e.g. Azulfidine RA®, Pleon RA®), Hydroxychloroquine (e.g. Quensyl®); Azathioprin, Methotrexate (e.g. Lantarel®, Metex®), Etanercept (Enbrel®), Adalimumab (Humira®), Infliximab (Remicade®), Tocilizumab (RoActemra®), Golimumab (Simponi®), Certolizumab (Cimzia®), Abatacept (Orencia®) for 6 months and if they are still in remission therapy will be discontinued.

SUMMARY:
This is a phase 3, multicenter, randomized, open, prospective, controlled, parallel-group intervention study in 318 patients with Rheumatoid Arthritis. The study is composed of 3 phases: a pre-randomization phase for up to 10 days followed by a 1-year randomized, open three arm treatment phase for each patient, followed by a 5-year observational phase for all patients still in remission.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is characterized by progressive synovitis leading to degradation of articular cartilage leading to erosions in juxtaarticular bones driven by auto antibodies. Few clinical studies could show that quick and thorough control of inflammatory processes could stop degradation processes [17, 18, 19, 20, 21] and had presumably better prognosis of remission than untreated and/or uncontrolled RA disease [20]. These studies aimed at low disease activity [20], often focused on early RA [18, 19], evaluating different therapy strategies, mostly escalating instead of deescalating medications [20, 21]. Real "RA- in - remission" or therapy reduction studies are missing up to now, even if first small trials focusing on one preparation showed promising results [16, 17].

In this study all conventional medications in usual combinations are being evaluated for the treatment of Rheumatoid Arthritis in different stages of disease duration. The study is scheduled as a 365-day (12-months), phase 3 multicenter, randomized, open, prospective, controlled, parallel-group intervention study in 318 patients with Rheumatoid Arthritis.

Based on the results of the clinical studies mentioned above, and the need for a guideline with therapy proposals for RA- patients in remission all current preparations will be evaluated in subjects under the controlled setting of a clinical study. The information obtained from this study will assess the formulation of new guidelines regarding patients with Rheumatoid Arthritis in remission.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form including written consentfor data protection
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must be male or female and aged ≥ 18 years at time of consent
* Must have a diagnosis of RA according to ACR criteria [26] for at least 12 months
* Must have a DAS 28 score of less than 2.6 (means: remission) at randomization (documented in at least three subsequent controls for six months; compare figure three in the appendix for details)
* At screening-visit patients should have been treated without alterations of therapy for at least six months with one of the following therapies: (i) one or more of the following conventional DMARDS (with or without concomitant use of glucocorticoids): Methotrexate, Leflunomide, Ciclosporine A, Sulfasalazine, Azathioprine or Hydroxychloroquine, (ii) a combination of a conventional DMARD (Methotrexate, Leflunomide, Ciclosporine A, Sulfasalazine, Azathioprine or Hydroxychloroquine) with one of the following biologicals (with or without concomitant use of glucocorticoids): Infliximab, Adalimumab, Etanercept, Tocilizumab, Golimumab, Certolizumab, Abatacept, (iii) or one of the biologicals mentioned above without combination with a conventional DMARD. All of the aforementioned biologicals are also allowed in combination with glucocorticoids, (iv) monotherapy treatment with glucocorticoids (without any DMARD or biological treatment).

Exclusion Criteria:

* Treatment with Rituximab during the last 12 months before screening
* Intake of a daily dosage of more than 5mg Prednisolone - equivalent during the last 6 months before randomization; intraarticular injections of glucocorticoids do not represent an exclusion criteria
* Current treatment with other DMARDS (for example MMF or preparations still in development) than mentioned above
* Any anti-inflammatory or immunosuppressive therapy for other reasons than RA during the last 3 months before screening
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Any other rheumatological/immunological disease such as Psoriasis, Psoriatic Arthritis, SLE, PSS, MCTD, M. Bechterew, M. Behcet or M. Wegener. Should the respective diagnosis be confirmed after inclusion into the study the patient will leave the study and data is recorded via "unscheduled visit"- and follow-up form
* Florid autoimmune conditions such as autoimmune hepatitis or Hashimoto's disease while still under treatment
* Patients with a florid malignancy
* Participation in another phase 1-4 treatment study for RA
* Patients who are younger than 18 years or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 und Abs. 3 AMG)
* Pregnant or lactating female
* Females of childbearing potential (FCBP is a sexually mature female who 1. has not undergone a hysterectomy or bilateral oophorectomy, or 2. has not been postmenopausal for at least 24 consecutive months) have to use adequate forms of contraception with respect to standard treatment recommendations. However if there is suspicion of a pregnancy in spite of standard treatment recommendations a urine pregnancy test is to be carried out by the Investigator
* Also males must also use adequate forms of contraception
* Patients who possibly are dependent on the Principal Investigator or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2009-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects in each treatment group who are still in remission after 12 months (remission defined as DAS 28 < 2.6) reduction or even discontinuation in RA-patients after achievement of long lasting remission. | 12 months

SECONDARY OUTCOMES:
Proportion of subjects in each treatment group who are still in remission after 3, 6, 9 months (remission defined as DAS 28 < 2.6). | 12 months
Proportion of subjects in each treatment group who are still in remission after 3, 6, 9 months (remission defined according to Pinals - criteria) | 12months
Proportion of subjects in each treatment group with increased disease activity | 12 months
Proportion of adverse events (to be documented via "unscheduled visit"-sheet) | 12 months
DAS 28 after 3, 6, 9 and 12 months | 12 months
CRP after 3, 6, 9 and 12 months | 12 months
ESR after 3, 6, 9 and 12 months | 12 months
Swollen joint counts after 3, 6, 9 and 12 months | 12 months
Tender joint counts after 3, 6, 9 and 12 months | 12 months
Patient self assessment of pain (VAS) after 3, 6, 9 and 12 months | 12 months
Physician's and patient's assessment of global disease activity (VAS) after 3, 6, 9 and 12 months | 12 months
Duration of joint stiffness after 3, 6, 9 and 12 months | 12 months
HAQ (Health Assessment Questionnaire) after 3, 6, 9 and 12 months | 12 months
SF-36 (Short Form) Score after 3, 6, 9 and 12 months | 12 months
Coping-Questionnaire after 3, 6, 9 and 12 months | 12 months
PASS (patient acceptable symptom state) after 3, 6, 9 and 12 months | 12 months
WPAI:RA (Work Productivity and Activity Impairment Questionnaire) after 3, 6, 9, 12 months | 12 months
BDI - II (Beck-Depression Inventory) after 3, 6, 9 and 12 months | 12 months
Flare Questionnaire RA (German version): At time of potential flare | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, Prof. Dr. univ., Study Director — University Clinic Erlangen, Clinical Trial Unit, Department of Internal Medicine 3, Rheumatology & Immunology
Locations (12):
- Germany (12):
  - Asklepios Klinikum Bad Abbach, Bad Abbach
  - Rheumapraxis Manger, Bamberg
  - Rheumapraxis Bayreuth, Bayreuth
  - Schlosspark-Klinik, Berlin
  - Schwerpunktpraxis für Rheumatologie Burghausen, Burghausen
  - PGRN.de Praxisgemeinschaft Rheumatologie Nephrologie, Erlangen
  - Universitätsklinikum Heidelberg; Medizinische Klinik V, Heidelberg
  - Gemeinschaftspraxis Dres. Demary und von Hinüber, Hildesheim
  - Praxiszentrum St. Bonifatius, München
  - Praxis Professor Nüsslein, Nuremberg
  - Universitätsklinikum Tübingen; Zentrum für Interdisziplinäre Klinische Immunologie, Rheumatologie und Autoimmunerkrankungen - INDIRA, Tübingen
  - Medizinische Klinik 2 und Poliklinik, Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tascilar K, Hagen M, Kleyer A, Simon D, Reiser M, Hueber AJ, Manger B, Englbrecht M, Finzel S, Tony HP, Schuch F, Kleinert S, Wendler J, Ronneberger M, Figueiredo CP, Cobra JF, Feuchtenberger M, Fleck M, Manger K, Ochs W, Schmitt-Haendle M, Lorenz HM, Nuesslein H, Alten R, Kruger K, Henes J, Schett G, Rech J. Treatment tapering and stopping in patients with rheumatoid arthritis in stable remission (RETRO): a multicentre, randomised, controlled, open-label, phase 3 trial. Lancet Rheumatol. 2021 Nov;3(11):e767-e777. doi: 10.1016/S2665-9913(21)00220-4. Epub 2021 Oct 1. PMID 38297524